CLINICAL TRIAL: NCT03385525
Title: A Phase 1, Open-label, Fixed-sequence Study to Evaluate the Effect of UGT Inhibition by Valproic Acid on the Pharmacokinetics of BIIB074 in Healthy Subjects
Brief Title: Study to Evaluate the Effect of UGT Inhibition by Valproic Acid on the Pharmacokinetics of BIIB074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802HV109
Record Dates: First submitted 2017-10-13; First posted 2017-12-28 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Drug Interaction
Keywords: Healthy Volunteer
MeSH Terms: interventions — vixotrigine; Valproic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BIIB074 150 mg and Valproic Acid 500 mg (Experimental): Participants will receive BIIB074 in tablet form in 150 mg doses. BIIB074 will be taken once daily (QD) on Days 1-16 after an 8-hour fast. Valproic Acid will be given in capsule form in 500 mg doses on prescription (TID) every 8 hours on Days 8-22. The morning dose on Day 16 will be coadministered with BIIB074 following an 8-hour fast.
  Interventions: Drug: BIIB074; Drug: Valproic Acid

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
Drug: Valproic Acid — Administered as specified in the treatment arm
  Other Names: Depakote, Depakene, Stavzor, and Valproic

SUMMARY:
The primary objective of this study is to evaluate the effect of multiple doses of the UGT inhibitor valproic acid on the single-dose pharmacokinetics of BIIB074. The secondary objectives of this study are to evaluate the safety and tolerability of BIIB074 when administered alone and when coadministered with the UGT inhibitor valproic acid and to evaluate the effect of the UGT inhibitor valproic acid on the PK of the M13, M14, and M16 metabolites of BIIB074.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body mass index between 18 and 32 kg/m^2, inclusive.
* Must be male, postmenopausal female, or surgically sterile female
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal (GI), hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening or Day -1
* History of, or positive test result at Screening for, human immunodeficiency virus (HIV)
* Treatment with any prescription or over-the-counter oral medication (excluding acetaminophen) within 14 days prior to Day -1 and an unwillingness or inability to refrain from this treatment during study participation, unless specifically permitted elsewhere within this protocol.
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Area Under the Concentration-Time Curve from Time Zero to Time of the Last Measurable Concentration (AUClast) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Time to Reach Maximum Observed Concentration (Tmax) for BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Time of Last Measured Serum Concentration (Tlast) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Elimination Half-Life (T 1/2) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Apparent Clearance (CL/F) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23
Apparent Volume of Distribution (V/F) of BIIB074 | Day 1 through Day 8, Day 16 through Day 23

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 32
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change from Baseline of Electrocardiogram (ECG) up to Day 23 | Day 1, 3, 8, 13, 16, 18, 23
Number of Participants with Abnormal Change from Baseline of Clinical Laboratory Parameters up to Day 23 | Day 3, 8, 13, 16, 18, 23
Number of Participants with Abnormal Change from Baseline of Vital Signs up to Day 23 | Day 1, 3, 8, 13, 16, 18, 23
Cmax of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
AUCinf of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
AUClast of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
Tmax of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
Tlast of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
T1/2 of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
Metabolite-to-Parent Ratio in AUC (MRauc) of BIIB074 Metabolites M13, M14, and M16 | Day 1 through Day 8, Day 16 through Day 23
Number of Participants with Abnormal Change from Baseline in Columbia Suicide Severity Rating (C-SSRS) scale | Day 8, 23, and once between Day 29-32
  C-SSRS is a suicidal ideation rating used to evaluate suicidality in children ages 12 and up. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Dallas, Texas, United States

REFERENCES:
- [Derived] Zhao Y, Kotecha M, Finnigan H, Serenko M, Naik H. Evaluation of the Effect of Uridine Diphosphate-Glucuronosyltransferases (UGT) Inhibition by Valproic Acid on Vixotrigine Pharmacokinetics in Healthy Volunteers. Clin Drug Investig. 2022 Oct;42(10):829-837. doi: 10.1007/s40261-022-01194-y. Epub 2022 Aug 31. PMID 36045316